CLINICAL TRIAL: NCT01114685
Title: Bone Mineral Density (BMD) Changes in a Bone Health Plan Using Two Versions of a Bone Health Supplement: A Comparative Effectiveness Research (CER) Study
Brief Title: A Comparison of Changes in Bone Density With the Same Bone-health Plan, But With Different Bone-health Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integrative Health Technologies, Inc. (Network)
Collaborators: AlgaeCal Inc. (Industry)
Responsible Party: Gilbert R. Kaats, PhD, Integrative Health Technologies, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AlgaeCal 1 & 2
Record Dates: First submitted 2010-04-19; First posted 2010-05-03 (Estimated); Last update posted 2010-05-03 (Estimated); Status verified 2010-04

CONDITIONS: Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Effects of taking AlgaeCal-1 (Active Comparator): Following a bone health plan with Algae-cal-1 supplement
  Interventions: Dietary Supplement: AlgaeCal-1
- Effects of taking AlgaeCal-2 (Active Comparator): Following a bone-health plan while consuming AlgaeCal 2
  Interventions: Dietary Supplement: AlgaeCal-2

INTERVENTIONS:
Dietary Supplement: AlgaeCal-1 — Daily consumption of 7 capsules containing bone health ingredients
  Arms: Effects of taking AlgaeCal-1
Dietary Supplement: AlgaeCal-2 — Taking 7 capsules a day for six months
  Arms: Effects of taking AlgaeCal-2

SUMMARY:
A comparison of changes in bone density following the same bone-health plan, but with a different bone-health supplement.

DETAILED DESCRIPTION:
The US Surgeon General's Report on Bone Health suggests America's bone-health is in jeopardy and issued a "call to action" to develop bone-health plans that:

1. improve nutrition,
2. increase health literacy and,
3. increase physical activity.

The purpose of this study was to use a comparative effective research model to compare 6-month changes in bone mineral density (BMD)in two study groups. Both followed the same bone health plan that contained the three components listed above with the same plant-source calcium supplement, but enhanced with different levels of calcium, vitamin D3, vitamin K and magnesium.

ELIGIBILITY:
Inclusion Criteria:

* All subjects were required to contact the physicians to ensure they had no medical issues that would preclude their participation.

Exclusion Criteria:

* Younger the 18 years of age, and
* Recommendations not to participate from their physicians.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2006-06; Primary Completion 2008-07 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Changes in Bone Mineral Density (BMD) | baseline and 6 months
  Measurements of bone mineral density were conducted at baseline and 6 months from baseline in two different study groups following the same bone-health behavior modification plan, but with different versions of a bone-health calcium supplement.

SECONDARY OUTCOMES:
A comparison of changes from baseline in 43-blood chemistry panel and a self-reported quality of life inventory in both study groups | six months
  Study subjects in both arms of the study completed a fasting 43-blood chemistry panel and an 84-item self-reported quality of life inventory at baseline and again after participating in the study for six months. No significant differences were found in the within-group changes from baseline or between the groups on both sets of measures.

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert R Kaats, PhD, Principal Investigator — Integrative Health Technologies; Harry G Preuss, MD, Principal Investigator — Georgetown University
Locations (1):
- Integrative Health Technologies, San Antonio, Texas, United States

REFERENCES:
- [Derived] Michalek JE, Preuss HG, Croft HA, Keith PL, Keith SC, Dapilmoto M, Perricone NV, Leckie RB, Kaats GR. Changes in total body bone mineral density following a common bone health plan with two versions of a unique bone health supplement: a comparative effectiveness research study. Nutr J. 2011 Apr 14;10:32. doi: 10.1186/1475-2891-10-32. PMID 21492428